CLINICAL TRIAL: NCT00003499
Title: Phase II Study of Antineoplaston A10 and AS2-1 in Patients With Non-Hodgkin's Lymphoma Low Grade
Brief Title: Antineoplaston Therapy in Treating Patients With Low-Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066538; BC-LY-6 (Other: BRI)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Low-Grade Lymphoma
Keywords: Low-grade non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with Low-grade non-Hodgkin's lymphoma will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)ANP

SUMMARY:
Current therapies for Low-grade Non-Hodgkin's Lymphoma provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Low-grade Non-Hodgkin's Lymphoma.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Low-grade Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
Low-grade Non-Hodgkin's Lymphoma patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Low-grade Non-Hodgkin's Lymphoma, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Low-grade Non-Hodgkin's Lymphoma.
* To determine objective response, tumor size is measured utilizing physical examination, radiologic studies, and bone marrow biopsies as necessary, performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage II, III, or IV low grade non-Hodgkin's lymphoma that is unlikely to respond to existing therapy or for which no established therapy exists NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC greater than 2,000/mm^3
* Platelet count greater than 20,000/mm^3

Hepatic:

* Bilirubin normal

Renal:

* Creatinine normal
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study
* No serious active infections

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since immunotherapy and recovered
* No concurrent immunomodulating agents (e.g., interferon, interleukin-2)

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered

Endocrine therapy:

* At least 4 weeks since prior corticosteroids
* No concurrent corticosteroids

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No prior antineoplaston therapy
* No other concurrent antineoplastic agents
* No concurrent antibiotics, antifungals, or antivirals

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 1996-03-06 (Actual); Primary Completion 2003-09-13 (Actual); Study Completion 2003-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-one patients were recruited between March 1996 and November 2002. All study subjects were seen at the Burzynski Clinic in Houston TX
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Patients with Low-grade non-Hodgkin's lymphoma will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 31
Completed | 23
Not Completed | 8
Not completed — Not evaluable | 8

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: Years] | 54.2 [37.1 to 69.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per The International Working Group response criteria (1999): Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 23
Participants
  Complete Response | 1
  Partial Response | 2
  Stable Disease | 14
  Progressive Disease | 6

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 31
Percentage of Participants
  6 months overall survival | 29
  12 months overall survival | 28
  24 months overall survival | 21
  36 months overall survival | 17
  48 months overall survival | 14
  60 months overall survival | 11

ADVERSE EVENTS:
Time Frame: 6 years, 8 months
Description: Adverse event data was collected through regular patient assessment and regular laboratory testing
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 10/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=31)
Hemoglobin (Blood and lymphatic system disorders) | 1 — The hemoglobin was not related to Antineoplaston therapy.
Left ventricular systolic dysfunction (Cardiac disorders) | 1 — The Left ventricular systolic dysfunction was not related to Antineoplaston therapy.
Infection (documented clinically): Blood (Infections and infestations) | 3 — The Infections (documented clinically): Blood werenot related to Antineoplaston therapy.
Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 2 — The Lung (pneumonias) were not related to Antineoplaston therapy.
Seizure (Nervous system disorders) | 1 — The Seizure was not related to Antineoplaston therapy.
Pain: Oral cavity (General disorders) | 1 — The Pain: Oral cavity was not related to Antineoplaston therapy.
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 — The Dyspnea (shortness of breath) was not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=31)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 10
Tinnitus (Ear and labyrinth disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 7
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 2
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3
Platelets (Blood and lymphatic system disorders) | 4
Cardiac Arrhythmia (Cardiac disorders) | 5
Central venous catheter infection (General disorders) | 2
Central venous catheter - non-functional (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 20
Fever (General disorders) | 5
Rigors/chills (General disorders) | 5
Hyperepidermisation (Skin and subcutaneous tissue disorders) | 2
Edema (General disorders) | 16
Diarrhea (Gastrointestinal disorders) | 8
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 22
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 10
Hemorrhage, GU (Renal and urinary disorders) | 2
Infection (documented clinically): Blood (Infections and infestations) | 6
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 2
Lung (pneumonia) (Infections and infestations) | 3
Mucosa (Infections and infestations) | 3
Skin (Infections and infestations) | 5
Upper airway (Infections and infestations) | 8
Alkaline phosphatase (Investigations) | 2
Hyperbilirubinemia (Investigations) | 3
Hyperglycemia (Investigations) | 5
Hypernatremia (Investigations) | 22
Hypocalcemia (Investigations) | 4
Hypochloremia (Investigations) | 2
Hypoglycemia (Investigations) | 3
Hypokalemia (Investigations) | 22
Hypomagnesemia (Investigations) | 2
SGOT (Investigations) | 8
SGPT (Investigations) | 4
Confusion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 9
Mood alteration (Nervous system disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 2
Somnolence/depressed level of consciousness (Nervous system disorders) | 9
Speech impairment (Nervous system disorders) | 2
Pain: Head/headache (Nervous system disorders) | 10
Pain: Joint (Musculoskeletal and connective tissue disorders) | 9
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No